CLINICAL TRIAL: NCT03090633
Title: Study of Fetoscopic Repair of Myelomeningocele in Fetuses With Isolated Spina Bifida
Brief Title: Fetoscopic Repair of Isolated Fetal Spina Bifida
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00123834
Record Dates: First submitted 2017-03-06; First posted 2017-03-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Spina Bifida; Myelomeningocele; Chiari Malformation Type 2; Neural Tube Defects; Spinal Dysraphism; Congenital Abnormality
Keywords: Fetoscopy; Fetal surgery; Fetal spina bifida
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele; Arnold-Chiari Malformation; Neural Tube Defects; Congenital Abnormalities | interventions — Fetoscopy

STUDY DESIGN:
Intervention Model Description: This is a single arm clinical study. All participants will undergo laparotomy with exteriorization of the uterus followed by minimally-invasive, fetoscopic repair of the fetal spina bifida lesion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fetoscopy (Experimental): All participants will undergo fetoscopic repair of fetal spina bifida.
  Interventions: Device: Fetoscopy

INTERVENTIONS:
Device: Fetoscopy — Minimally invasive in-utero surgery
  Other Names: Karl Storz Endoscopy America, Inc.; Richard Wolf Medical Instruments, Corp.; Cook Medical, Inc.; Pare Surgical, Inc.

SUMMARY:
The purpose of this investigation is to evaluate maternal and fetal outcomes following fetoscopic repair of fetal spina bifida at the Johns Hopkins Hospital.

The hypothesis of this study is that fetoscopic spina bifida repair is feasible and has the same effectiveness as open repair of fetal spina bifida, but with the benefit of significantly lower maternal and fetal complication rates. The fetal benefit of the procedure will be the prenatal repair of spina bifida. The maternal benefit of fetoscopic spina bifida repair will be the avoidance of a large uterine incision. This type of incision increases the risk of uterine rupture and requires that all future deliveries are by cesarean section. The use of the minimally invasive fetoscopic surgical technique may also lower the risk of preterm premature rupture of membranes and preterm birth compared to open fetal surgery. Finally, successful fetoscopic spina bifida repair also makes vaginal delivery possible.

DETAILED DESCRIPTION:
Spina bifida is a congenital anomaly that results from incomplete closure of the neural tube between 22 and 28 embryological days. Its incidence is approximately 2-4 cases per 10,000 births, and it is considered the most common congenital central nervous system anomaly that is compatible with life (CDC). Open spina bifida can present as a flat defect without a covering (myeloschisis), it may have a membranous covering (meningocele), or the fluid may be extruded into a fluid filled sac (myelomeningocele or MMC). Spina bifida can lead to lifelong sequelae that are the result of additional insult to the nervous system that occurs during fetal life as a consequence of the anomaly in the spinal cord. Downward displacement of the brain stem results in hindbrain herniation and the Chiari II malformation during fetal life leading to non-communicating hydrocephalus. Concurrently, intrauterine injury to exposed neural elements leads to neurologic dysfunction.

Despite improved care and technology, 2-year survival of affected individuals is 75%. The need for ventriculoperitoneal shunting for hydrocephaly is related to the level of the lesion and ranges between 88-97% for thoracolumbar lesions. Shunt placement in and of itself is associated with complications such as obstruction, infection, and displacement requiring repeated shunt revisions as early as the first year of life. The majority (75%) of patients with hydrocephaly have radiologic evidence of the Arnold-Chiari II malformation (hindbrain herniation, brain stem abnormalities, and small posterior fossa), which are associated with symptoms of apnea, swallowing difficulties, quadriparesis, balance issues, and coordination difficulties. The lesion level also correlates to the functional motor level; in general, the rate of being wheelchair-bound increases from 17% in sacral lesions to 90% of patients with a thoracic level lesions. Almost 90% of infants with spina bifida require intervention for a foot deformity to allow weight bearing activities. Bowel and urinary tract complications are common, and while children with spina bifida can achieve normal intelligence, they are at risk for neurocognitive and language difficulties that might impact school performance and the ability to live independently. The acquired disabilities tend to increase into adulthood and are attributed to a high rate of unexpected death. Overall, the most frequent form of spina bifida is MMC associated with hydrocephaly, lower limb paralysis, and bowel and bladder dysfunction.

The ultimate neurologic deficit that occurs with MMC that is established at birth is thought to originate from two mechanisms. First, there is an anatomic abnormality of a relatively normal spinal cord that then becomes secondarily damaged by the intrauterine environment through amniotic fluid exposure, direct trauma, hydrodynamic pressure, or a combination of these. This "two-hit hypothesis" is based on the observation that progressive neurologic damage develops in fetuses with MMC as gestation advances and results in irreversible neurologic damage at birth. The potential ability to ameliorate secondary damage caused by exposure to the in utero environment gave rise to the concept of fetal surgery for MMC repair.

The prenatal diagnosis of MMC with Chiari II malformation can be determined by ultrasound in almost all cases between 14-20 weeks gestation, and in the second trimester diagnosis is 97% sensitive and 100% specific. Accordingly, potential candidates for prenatal repair can be identified early in pregnancy leaving adequate time for detailed anatomic evaluation, genetic workup, and multidisciplinary patient counseling.

Because of the lifelong morbidity associated with the condition and the ability to accurately make a prenatal diagnosis of spina bifida, the idea of in-utero surgery to improve outcomes was conceived. Early animal studies and subsequent human pilot studies laid the groundwork for the Management of Myelomeningocele Study (MOMS trial). While the animal models supported the concept of the two-hit theory and the principle of improved neurologic function after in utero repair, these findings could not be directly extrapolated to human application. The National Institutes of Health (NIH) sponsored the multicenter randomized MOMS trial that compared outcomes between prenatal MMC repair with standard postnatal management. Prenatal MMC repair was performed between 19-25 6/7 weeks gestational age. The fetal repair involves a two to three layer closure similar to neonatal surgery. The neural placode is sharply dissected from the surrounding tissue. The dura and myofascial flaps are then re-approximated over the neural placode. A running suture is then used to close the skin. The coverage must be completely "water tight" to prevent the leakage of cerebrospinal fluid through the MMC defect that leads to hindbrain herniation in order to prevent amniotic fluid exposure which damages the neural tissues in the MMC defect. The uterus was closed in two layers (running closure and interrupted stay sutures) and then covered with an omental flap. Following prenatal MMC repair, patients remained near the fetal surgery center until delivery by cesarean section.

The study demonstrated that prenatal MMC repair was associated with a significantly lower rate of shunting, and hindbrain herniation and produced better motor outcomes. In the prenatal surgery group, functional motor level was better by two or more levels from anatomic level in 32% and better by one level in 11% compared with 12% and 9%, respectively.

The major risks of prenatal surgery for the fetus include chorioamniotic membrane separation (26% vs. 0%, p < 0.001), spontaneous rupture of membranes (46 vs. 8% p < 0.001), and spontaneous preterm labor with preterm birth (38 vs. 14%, p<0.001). This led to the lower gestational age at delivery in the prenatal surgery group of 34 weeks compared with 37 weeks in the postnatal surgery group (p < 0.001). Within the prenatal surgery group, 13% of patients delivered at a severely premature gestation of < 30 weeks and 33% at 30-34 weeks.

Prenatal MMC repair is associated with significant maternal risks, including pulmonary edema (6%) and blood transfusion at delivery (9%). Hysterotomy thinning was observed in 25% of women and uterine dehiscence and 1% of women. Moreover, women have a 14% risk for scar dehiscence in future pregnancies and invariably require delivery by cesarean section. The reason for the increased incidence of these complications is related to the nature of the open fetal procedure, which involves a multi-faceted invasive approach including maternal laparotomy, large hysterotomy with uterine edge stapling, and open fetal repair of the spina bifida defect that may involve manipulation and exposure of the fetus for a significant amount of time. Nevertheless, the MOMS trial demonstrated significant fetal and neonatal benefit. While maternal risks remain significant, prenatal MMC repair has been adopted as an accepted care standard across the United States.

Fetal endoscopic surgery has progressed rapidly over the past few decades and many fetal therapy centers are now able to perform a number of intricate procedures inside the uterus. Since fetoscopy offers a less invasive therapeutic option than open fetal surgery, there have been several efforts to develop this technique for MMC repair with the goal to duplicate the beneficial fetal effects while avoiding the significant maternal morbidity. Animal and human experimental experience with fetoscopic repair of MMC has been reported, showing the feasibility of covering the defect with a patch, sealant, or by full repair. These fetoscopic repairs are typically performed using at least two ports. Due to the complex surgical manipulations, particularly when patch closures are performed, operative times are long and are associated with significant obstetric morbidities.

A maneuver associated with improved ability to perform a fetoscopic repair is intrauterine insufflation with carbon dioxide. This provides a dry working area for the surgeon to perform the closure. The fetal therapy team at the Johns Hopkins Center for Fetal Therapy has previously utilized intrauterine carbon dioxide (CO2) insufflation in situations where a dry surgical environment was required. Most recently a two port-technique for fetoscopic MMC repair under CO2 insufflation was described by the Baylor College of Medicine/Texas Children's Fetal Center using the externalized approach. This technique employs a laparotomy to exteriorize the uterus, which can then be positioned for access with two surgical ports regardless of the placental location. After CO2 insufflation and fetal anesthesia is administered, the MMC repair is performed after sharp dissection of the placode using a mattress suture. This approach is designed to decrease the maternal obstetric risks while preserving the fetal benefits.

The technique employs low-pressure uterine CO2 distention at 8-12 mmHg. In addition, significantly quicker neural tube repair is possible because of improved access to the fetus, ability to manipulate the fetus into the required position, and superior port placement resulting from the exteriorized maternal uterus. As a result only two ports are required and these can be sutured into the uterus allowing a closed seal and minimizing gas leakage. Finally, recent advances in small diameter surgical instruments (Storz 1.5 - 3mm surgical sets) allow a full surgical repair to be performed via a fetoscopic approach.

The purpose of the current study is to evaluate the feasibility of performing fetoscopic spina bifida repair at Johns Hopkins Hospital and the fetal and maternal outcomes following this approach.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years and older who are able to consent
* Singleton pregnancy
* Normal fetal karyotype
* Isolated fetal spina bifida with the upper lesion level between T1-S1
* Gestational age between 19+0 to 25+6 weeks gestation

Exclusion Criteria:

* Pregnant women less than 18 years of age
* Multiple gestation
* Fetal anomaly unrelated to spina bifida
* Maternal contraindication to fetoscopic surgery
* Severe maternal medical condition in pregnancy
* Technical limitations preluding fetoscopic surgery
* Preterm labor
* Cervical length < 25mm
* Placenta previa
* Psychosocial ineligibility precluding consent
* Maternal Beck Depression Inventory score ≥ 17

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a study of pregnant women.
Enrollment: 30 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Ability to perform fetoscopic spina bifida repair | From time of surgery until delivery (up to 21 weeks)
  Successful complete closure of the defect fetoscopically and reversal of hindbrain herniation on ultrasound and MRI prior to delivery

SECONDARY OUTCOMES:
Maternal obstetric outcome as evidenced by preterm premature rupture of membranes | From time of surgery until 37 weeks of gestation (up to 18 weeks)
  Preterm premature rupture of membranes occuring any time from surgery until 37 weeks of gestation
Maternal obstetric outcome as evidenced by preterm labor leading to delivery at less than 34 weeks of gestation | From time of surgery until 34 weeks of gestation (up to 15 weeks)
  Preterm labor occuring at any time from surgery leading to delivery before 34 weeks of gestation
Maternal obstetric outcome as evidenced by gestational age at delivery | From time of surgery until delivery (up to 21 weeks)
  Gestational age of delivery regardless of indication
Maternal obstetric outcome as evidenced by the ability to delivery vaginally | From time of surgery until delivery (up to 21 weeks)
  Mode of delivery - either vaginal or cesarean section
Adverse fetal or neonatal outcome as evidenced by fetal or neonatal death | From the time of surgery until 28 days of life (up 25 weeks)
  Composite of fetal or neonatal death
Adverse early childhood outcome as evidenced by need for a cerebrospinal fluid shunt | From the time of birth until 12 months of life
  Need for a cerebrospinal fluid shunt within the first year of life
Neurodevelopmental outcome as evaluated by the Bayley Scales of Infant Development II | 30 months of age
  Score of the Mental Developmental Index of the Bayley Scales of Infant Development II at 30 months of age. The score ranges from 50 (minimum) to 150 (maximum). A score of <70 indicates severe developmental delay; 70-84 indicates moderate delay; >85 indicates no delay.
Early childhood motor function on physical examination | 30 months of age
  Difference between the anatomic upper border of the lesion level and motor function based on the physical examination at 30 months of age. A positive score of 2 indicates a functional level 2 vertebrae higher than lesion level. A score of -2 indicates a function level 2 vertebrae lower than the lesion level.

CONTACTS AND LOCATIONS:
Overall Officials: Jena Miller, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Collaborate in the International Fetoscopic Neural Tube Defect (NTD) Consortium - A Limited Data Set will be entered into a website maintained by Baylor College of Medicine. The data will be combined with data provided by other members of the Consortium to provide a comprehensive Data Base that will be accessible by all Consortium members.
Time Frame: After execution of the Consortium and Data Base Provider Agreement, PROVIDER shall enter the Limited Data Set to the website maintained by BAYLOR. This Agreement shall terminate when all of the Limited Data Set provided by PROVIDER to BAYLOR for the Permitted Data Use is destroyed.
Access Criteria: The Data Base will be accessible by all Consortium members.

REFERENCES:
- [Background] Bowman RM, McLone DG, Grant JA, Tomita T, Ito JA. Spina bifida outcome: a 25-year prospective. Pediatr Neurosurg. 2001 Mar;34(3):114-20. doi: 10.1159/000056005. PMID 11359098
- [Background] Caldarelli M, Di Rocco C, La Marca F. Shunt complications in the first postoperative year in children with meningomyelocele. Childs Nerv Syst. 1996 Dec;12(12):748-54. doi: 10.1007/BF00261592. PMID 9118142
- [Background] Cass AS, Luxenberg M, Johnson CF, Gleich P. Incidence of urinary tract complications with myelomeningocele. Urology. 1985 Apr;25(4):374-8. doi: 10.1016/0090-4295(85)90492-3. PMID 3984125
- [Background] Cochrane DD, Wilson RD, Steinbok P, Farquharson DF, Irwin B, Irvine B, Chambers K. Prenatal spinal evaluation and functional outcome of patients born with myelomeningocele: information for improved prenatal counselling and outcome prediction. Fetal Diagn Ther. 1996 May-Jun;11(3):159-68. doi: 10.1159/000264297. PMID 8739582
- [Background] Centers for Disease Control and Prevention (CDC). Hospital stays, hospital charges, and in-hospital deaths among infants with selected birth defects--United States, 2003. MMWR Morb Mortal Wkly Rep. 2007 Jan 19;56(2):25-9. PMID 17230142
- [Background] Fontecha CG, Peiro JL, Sevilla JJ, Aguirre M, Soldado F, Fresno L, Fonseca C, Chacaltana A, Martinez V. Fetoscopic coverage of experimental myelomeningocele in sheep using a patch with surgical sealant. Eur J Obstet Gynecol Reprod Biol. 2011 Jun;156(2):171-6. doi: 10.1016/j.ejogrb.2010.12.046. Epub 2011 Feb 25. PMID 21353374
- [Background] Hutchins GM, Meuli M, Meuli-Simmen C, Jordan MA, Heffez DS, Blakemore KJ. Acquired spinal cord injury in human fetuses with myelomeningocele. Pediatr Pathol Lab Med. 1996 Sep-Oct;16(5):701-12. PMID 9025869
- [Background] Just M, Schwarz M, Ludwig B, Ermert J, Thelen M. Cerebral and spinal MR-findings in patients with postrepair myelomeningocele. Pediatr Radiol. 1990;20(4):262-6. doi: 10.1007/BF02019662. PMID 2336286
- [Background] Kohl T, Tchatcheva K, Weinbach J, Hering R, Kozlowski P, Stressig R, Gembruch U. Partial amniotic carbon dioxide insufflation (PACI) during minimally invasive fetoscopic surgery: early clinical experience in humans. Surg Endosc. 2010 Feb;24(2):432-44. doi: 10.1007/s00464-009-0579-z. Epub 2009 Jun 30. PMID 19565298
- [Background] Kohl T, Tchatcheva K, Merz W, Wartenberg HC, Heep A, Muller A, Franz A, Stressig R, Willinek W, Gembruch U. Percutaneous fetoscopic patch closure of human spina bifida aperta: advances in fetal surgical techniques may obviate the need for early postnatal neurosurgical intervention. Surg Endosc. 2009 Apr;23(4):890-5. doi: 10.1007/s00464-008-0153-0. Epub 2008 Sep 26. PMID 18818968
- [Background] Meuli M, Meuli-Simmen C, Hutchins GM, Seller MJ, Harrison MR, Adzick NS. The spinal cord lesion in human fetuses with myelomeningocele: implications for fetal surgery. J Pediatr Surg. 1997 Mar;32(3):448-52. doi: 10.1016/s0022-3468(97)90603-5. PMID 9094015
- [Background] Mitchell LE, Adzick NS, Melchionne J, Pasquariello PS, Sutton LN, Whitehead AS. Spina bifida. Lancet. 2004 Nov 20-26;364(9448):1885-95. doi: 10.1016/S0140-6736(04)17445-X. PMID 15555669
- [Background] Oakeshott P, Hunt GM, Poulton A, Reid F. Expectation of life and unexpected death in open spina bifida: a 40-year complete, non-selective, longitudinal cohort study. Dev Med Child Neurol. 2010 Aug;52(8):749-53. doi: 10.1111/j.1469-8749.2009.03543.x. Epub 2009 Dec 9. PMID 20015251
- [Background] Oakeshott P, Hunt GM. Long-term outcome in open spina bifida. Br J Gen Pract. 2003 Aug;53(493):632-6. PMID 14601340
- [Background] Pedreira DA, Oliveira RC, Valente PR, Abou-Jamra RC, Araujo A, Saldiva PH. Gasless fetoscopy: a new approach to endoscopic closure of a lumbar skin defect in fetal sheep. Fetal Diagn Ther. 2008;23(4):293-8. doi: 10.1159/000123616. Epub 2008 Apr 14. PMID 18417995
- [Background] Peiro JL, Fontecha CG, Ruano R, Esteves M, Fonseca C, Marotta M, Haeri S, Belfort MA. Single-Access Fetal Endoscopy (SAFE) for myelomeningocele in sheep model I: amniotic carbon dioxide gas approach. Surg Endosc. 2013 Oct;27(10):3835-40. doi: 10.1007/s00464-013-2984-6. Epub 2013 May 14. PMID 23670742
- [Background] Rintoul NE, Sutton LN, Hubbard AM, Cohen B, Melchionni J, Pasquariello PS, Adzick NS. A new look at myelomeningoceles: functional level, vertebral level, shunting, and the implications for fetal intervention. Pediatrics. 2002 Mar;109(3):409-13. doi: 10.1542/peds.109.3.409. PMID 11875133
- [Background] Shin M, Kucik JE, Siffel C, Lu C, Shaw GM, Canfield MA, Correa A. Improved survival among children with spina bifida in the United States. J Pediatr. 2012 Dec;161(6):1132-7. doi: 10.1016/j.jpeds.2012.05.040. Epub 2012 Jun 23. PMID 22727874
- [Background] Vachha B, Adams R. Language differences in young children with myelomeningocele and shunted hydrocephalus. Pediatr Neurosurg. 2003 Oct;39(4):184-9. doi: 10.1159/000072469. PMID 12944698
- [Background] Verbeek RJ, Heep A, Maurits NM, Cremer R, Hoving EW, Brouwer OF, van der Hoeven JH, Sival DA. Fetal endoscopic myelomeningocele closure preserves segmental neurological function. Dev Med Child Neurol. 2012 Jan;54(1):15-22. doi: 10.1111/j.1469-8749.2011.04148.x. Epub 2011 Nov 29. PMID 22126123
- [Background] Wilson RD, Lemerand K, Johnson MP, Flake AW, Bebbington M, Hedrick HL, Adzick NS. Reproductive outcomes in subsequent pregnancies after a pregnancy complicated by open maternal-fetal surgery (1996-2007). Am J Obstet Gynecol. 2010 Sep;203(3):209.e1-6. doi: 10.1016/j.ajog.2010.03.029. PMID 20537307
- [Background] Lavigne JV, Faier-Routman J. Psychological adjustment to pediatric physical disorders: a meta-analytic review. J Pediatr Psychol. 1992 Apr;17(2):133-57. doi: 10.1093/jpepsy/17.2.133. PMID 1534367
- [Background] Lennon CA, Gray DL. Sensitivity and specificity of ultrasound for the detection of neural tube and ventral wall defects in a high-risk population. Obstet Gynecol. 1999 Oct;94(4):562-6. doi: 10.1016/s0029-7844(99)00399-3. PMID 10511359
- [Background] Northrup H, Volcik KA. Spina bifida and other neural tube defects. Curr Probl Pediatr. 2000 Nov-Dec;30(10):313-32. doi: 10.1067/mpp.2000.112052. PMID 11147289
- [Background] Baschat AA, Ahn ES, Murphy J, Miller JL. Fetal blood-gas values during fetoscopic myelomeningocele repair performed under carbon dioxide insufflation. Ultrasound Obstet Gynecol. 2018 Sep;52(3):400-402. doi: 10.1002/uog.19083. Epub 2018 Jul 18. PMID 29750436
- [Background] Miller JL, Ahn ES, Garcia JR, Miller GT, Satin AJ, Baschat AA. Ultrasound-based three-dimensional printed medical model for multispecialty team surgical rehearsal prior to fetoscopic myelomeningocele repair. Ultrasound Obstet Gynecol. 2018 Jun;51(6):836-837. doi: 10.1002/uog.18891. No abstract available. PMID 28850758
- [Background] Belfort MA, Whitehead WE, Shamshirsaz AA, Bateni ZH, Olutoye OO, Olutoye OA, Mann DG, Espinoza J, Williams E, Lee TC, Keswani SG, Ayres N, Cassady CI, Mehollin-Ray AR, Sanz Cortes M, Carreras E, Peiro JL, Ruano R, Cass DL. Fetoscopic Open Neural Tube Defect Repair: Development and Refinement of a Two-Port, Carbon Dioxide Insufflation Technique. Obstet Gynecol. 2017 Apr;129(4):734-743. doi: 10.1097/AOG.0000000000001941. PMID 28277363
- [Background] Kohl T, Ziemann M, Weinbach J, Tchatcheva K, Gembruch U, Hasselblatt M. Partial amniotic carbon dioxide insufflation during minimally invasive fetoscopic interventions seems safe for the fetal brain in sheep. J Laparoendosc Adv Surg Tech A. 2010 Sep;20(7):651-3. doi: 10.1089/lap.2010.0068. PMID 20822417
- [Background] Pedreira DA, Zanon N, Nishikuni K, Moreira de Sa RA, Acacio GL, Chmait RH, Kontopoulos EV, Quintero RA. Endoscopic surgery for the antenatal treatment of myelomeningocele: the CECAM trial. Am J Obstet Gynecol. 2016 Jan;214(1):111.e1-111.e11. doi: 10.1016/j.ajog.2015.09.065. Epub 2015 Sep 18. PMID 26386383
- [Background] Saiki Y, Litwin DE, Bigras JL, Waddell J, Konig A, Baik S, Navsarikar A, Rebeyka IM. Reducing the deleterious effects of intrauterine CO2 during fetoscopic surgery. J Surg Res. 1997 Apr;69(1):51-4. doi: 10.1006/jsre.1997.5026. PMID 9202646
- [Background] Zerris VA, James KS, Roberts JB, Bell E, Heilman CB. Repair of the dura mater with processed collagen devices. J Biomed Mater Res B Appl Biomater. 2007 Nov;83(2):580-8. doi: 10.1002/jbm.b.30831. PMID 17465025
- [Result] Adzick NS, Thom EA, Spong CY, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Dabrowiak ME, Sutton LN, Gupta N, Tulipan NB, D'Alton ME, Farmer DL; MOMS Investigators. A randomized trial of prenatal versus postnatal repair of myelomeningocele. N Engl J Med. 2011 Mar 17;364(11):993-1004. doi: 10.1056/NEJMoa1014379. Epub 2011 Feb 9. PMID 21306277
- [Result] Belfort MA, Whitehead WE, Shamshirsaz AA, Ruano R, Cass DL, Olutoye OO. Fetoscopic Repair of Meningomyelocele. Obstet Gynecol. 2015 Oct;126(4):881-884. doi: 10.1097/AOG.0000000000000835. PMID 25923030